CLINICAL TRIAL: NCT00378677
Title: Pilot Study of Cyclosporine A Dry Powder Inhalation in Lung Transplant Patients With Bronchiolitis Obliterans Syndrome
Brief Title: Dry Powder Inhalation of Cyclosporine A in Lung Transplant Patients With Bronchiolitis Obliterans Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSA-DPI
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Lung Transplantation; Bronchiolitis Obliterans
Keywords: Powder inhalation; Side effects; Nephrotoxicity; Calcineurin inhibitor; Bronchiolitis obliterans syndrome; Forced Expiratory Volume
MeSH Terms: conditions — Bronchiolitis Obliterans; Bronchiolitis Obliterans Syndrome | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Cyclosporine A dry powder inhalation (Drug)

SUMMARY:
The purpose of this study is to investigate whether dry powder inhalation of Cyclosporine A is beneficial in lung transplant patients with Bronchiolitis Obliterans Syndrome. For patients suffering from this syndrome often no therapeutic options are available. Furthermore, the side effects of the maintenance therapy leaves no room for dose increments. The hypothesis for this trial is that when Cyclosporine A is administered locally (in the lungs) chronic rejection can be treated more effectively without extra systemic side effects.

DETAILED DESCRIPTION:
Because calcineurin inhibitors are not completely effective in a full prevention of acute rejection and the corresponding chronic disfunction of the transplanted organ (Bronchiolitis Obliterans Syndrome, BOS) a rejection risc remains. To effectively treat BOS high doses of calcineurin inhibitors are necessary. On the other hand these high doses lead te serious side effects. The search for a balance between effectiveness and side effects leads to dose adjustments. Ultimately, chronic rejection is unstoppable.

In order to treat chronic rejection higher doses of calcineurin inhibitors are not a therapeutic option. The only option to reach a high dose in the target organ without extra systemic side effects would be inhalation. Indeed, this has been extensively investigated at the University of Pittsburgh (lead investigator Iacono).

The intervention in the Pittsburgh trials existed of nebulization of Cyclosporine in propylene glycol with pretreatment of nebulization of lidocaine/albuterol in order to make the inhalation tolerable.

The investigational drug in this trial consists of dry powder inhalation of a sugar-glass based solid dispersion containing cyclosporine A. The effectiveness is measured by comparing the Forced Expiratory Volume in 1 second (FEV1) before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Primary lung transplant
* Tacrolimus as maintenance therapy
* Bronchiolitis Obliterans Syndrome stages 1 - 3: FEV1<80% of baseline
* At least 3 months after last usual BOS intervention
* Declining FEV1 after last usual BOS intervention

Exclusion Criteria:

* Cyclosporine as maintenance therapy
* Bronchiolitis Obliterans Syndrome 0: FEV1>80%
* Renal failure: Glomerular Filtration Rate < 30 ml/min
* Chronic airway infections
* Clinical stability
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7
Dates: Start 2007-02

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 second before and after intervention
Amount of lung deposition of cyclosporine A
Systemic uptake of Cyclosporine A

SECONDARY OUTCOMES:
Kidney function (GFR and serum creat)

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Zijlstra, Pharmacist, Principal Investigator — University of Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands